CLINICAL TRIAL: NCT02591264
Title: Periprocedural Myocardial Infarction: the Role of Human Neutrophil Peptide-1 to 3
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 90-14-HYMC
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Coronary Thrombosis
MeSH Terms: conditions — Coronary Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood sample — Blood sample drawn from participants for analysis of neutrophil peptide level

SUMMARY:
The aim of this study is to determine the role of human neutrophil peptide-1 to 3 in the occurrence of periprocedural myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Troponin negative patients
* Stable angina
* Unstable angina
* Positive screening tests

Exclusion Criteria:

* Troponin positive
* Technical failure of procedure
* Hemodynamic unstability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Troponin negative patients assigned for stent implantation in our medical institution.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Human Neutrophil Peptide Level | Two hours
  Laboratory analysis and measurement of Human Neutrophil Peptide-1 to 3 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel